CLINICAL TRIAL: NCT02649010
Title: A Performance Evaluation of the Enlite 3 Sensor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP309
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Type 2 Diabetes; Enlite 3 Sensor; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Subjects will be randomly assigned to 2 groups (Group A & Group B) that will determine when they will be participating in the in-clinic YSI frequent sample testing.
  Interventions: Device: Enlite 3 Sensor
- Group B (Active Comparator): Subjects will be randomly assigned to 2 groups (Group A & Group B) that will determine when they will be participating in the in-clinic YSI frequent sample testing.
  Interventions: Device: Enlite 3 Sensor

INTERVENTIONS:
Device: Enlite 3 Sensor — Use of Enlite 3 Sensor over 168 hours (7 days) when inserted in the arm and used with the 640G Pump in subjects aged 14-75 years who have had a diagnosis of type 1 or type 2 diabetes for at least 12 months.

SUMMARY:
The purpose of this study is to support the use of the Enlite 3 sensor in arm and thigh in subjects age 14 - 75 years and provide additional characterization of the Enlite 3 sensor performance in arm in subjects age 14 - 75 years.

DETAILED DESCRIPTION:
The study is a multi-center, randomized, prospective single-sample correlational design without controls.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 14 - 75 years of age at time of screening.
2. A clinical diagnosis of type 1 or 2 diabetes for a minimum of 9 months duration as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Adequate venous access as assessed by investigator or appropriate staff
4. Subjects participating in the high and low glucose challenges must have an established insulin carbohydrate ratio(s) and insulin sensitivity ratio. (The term "established" refers to a ratio that has been previously defined and tested prior to screening visit). Subjects without established ratios may participate under observation only.

Exclusion Criteria:

1. Subject will not tolerate tape adhesive in the area of Enlite 3 Sensor placement as assessed by qualified individual.
2. Subject has any unresolved adverse skin condition in the area of Enlite 3 Sensors or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Subject is female and has a positive pregnancy screening test
5. Females of child bearing age and who are sexually active should be excluded if they are not using a form of contraception deemed reliable by investigator.
6. Subject is female and plans to become pregnant during the course of the study
7. Subject has had a hypoglycemic seizure within the past 6 months.
8. Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to screening visit.
9. Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to screening visit.
10. Subject has a history of a seizure disorder.
11. Subject has central nervous system or cardiac disorder resulting in syncope.
12. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease.
13. Subject has a hematocrit(Hct) lower than the normal reference range.
14. Subject has a history of adrenal insufficiency

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Enlite 3 Sensor inserted at Arm accuracy using a real time device: (640G pump) with the minimum calibration requirements (every 12 hours after the second calibration) will be evaluated. | 1 month
  Glucose sensor values will be compared to Yellow Spring Instruments (YSI)plasma glucose values during Frequent Sample Testing.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lee, MD, Study Director — Medtronic Diabetes
Locations (2):
- United States (2):
  - Diablo Clinical Research, Walnut Creek, California
  - Rainier Clinical Research Center, Renton, Washington